CLINICAL TRIAL: NCT01208363
Title: Improving Iron Status Through Consumption Of Iron Fortified Cowpea: An Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Noguchi Memorial Institute for Medical Research (Other); Nestlé Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COWPEA; WUR10/13 (Other: WUR10/13)
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-03

CONDITIONS: Anemia; Low Iron Stores
Keywords: Iron fortification; polyphenols; NaFeEDTA; cowpea; school feeding program
MeSH Terms: conditions — Anemia | interventions — Fe(III)-EDTA

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unfortified Toubani (No Intervention): Children in the school will receive, 3 times per week 66g of raw unfortified (no added Fe) cowpea in form of Toubani (a cowpea based snack).
  Interventions: Dietary Supplement: Cowpea fortified with NaFeEDTA, in form of Toubani.
- Fortified Cowpea (Active Comparator): Study subjects will receive 3 times per week, as part of the school feeding programme 66g of raw fortified cowpea (with added 10mg Fe as NaFeEDTA)in form of Toubani (a cowpea based snack).
  Interventions: Dietary Supplement: Cowpea fortified with NaFeEDTA, in form of Toubani.

INTERVENTIONS:
Dietary Supplement: Cowpea fortified with NaFeEDTA, in form of Toubani. — 66g raw Cowpea fortified with 10 mg Fe as NaFeEDTA, in form of Toubani, a cowpea snack. Ther snack will be given to the participants 3 times per week, for six month integrated in the school feeding trial.

SUMMARY:
Rationale: Iron deficiency and zinc deficiency, are of public health significance in sub-Saharan Africa. An estimated 50% of children (5-14 years) in developing countries suffer from anaemia, half of which is estimated iron deficiency anaemia. Interventions have been designed and implemented over the years towards solving hunger and anaemia especially among school age children. One of such interventions is School Feeding Programme (SFP) which is common in both developing and industrialized countries. SFP has been part of the Ghanaian educational system for well over 40 years, albeit on small scale. The main stay of the programme that makes it distinguishable from other past and existing school feeding programmes is its reliance on locally produced and available foods, such as cowpeas. Legume staples like cowpea have been identified to be important sources of protein and non-heme iron to rural populations of developing countries like Ghana. The problem however is the low bioavailability of these micronutrients from these legumes.

Objective: To assess the efficacy of iron fortified cowpea based meal (Tubani) in improving iron status of primary school children in rural northern Ghana Study design: A randomized double blind parallel design will be conducted. One group will receive iron fortified Tubani with NaFeEDTA and the other group will receive unfortified Tubani.

Study population: Two hundred and forty apparently healthy pupils in lower primary school will participate. The participating schools have a school feeding programme currently in operation.

Intervention (if applicable): Children will be fed Tubani containing 10mg of fortification iron (in the form of NaFeEDTA) three times in a week for six months. Weight, height and blood samples will be measured at baseline and after six months of intervention. Participants will be treated against intestinal parasites before start of intervention and halfway through the intervention.

Main study parameters/endpoints: The main study endpoint is iron-deficiency anaemia (IDA). IDA will be defined as concurrent anaemia and iron deficiency. Whole blood will be collected for the analysis of Hb, serum ferritin (SF), serum transferring receptor (sTfR) and C-reactive protein (CRP). Anemia will be defined as a hemoglobin concentration <115 g/L, and iron deficiency will be defined as an SF concentration <12 µg/L.

Venipunctures occasionally lead to bruises or small local inflammation which usually disappear within one week. To minimize this risk, blood collection will be performed by a trained and experienced phlebotomists. Written informed consent will be obtained from all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Children 6-12 years old
* Regularly attending school, in grades 1-3
* Apparently healthy, free of chronic illnesses and not taking chronic medication.
* No medication nor supplemental iron at time of entry into the study
* Informed consent obtained from at least one parent or guardian

Exclusion Criteria:

* Children with severe anemia (Hb<70 g/l).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-04 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Iron deficiency anemia, defined by Hb<115 g/l; SF<12 microgram/l | Duration will be 6 months. Measurements will be performed at start and after 6 months of intervention.
  Autcome parameters are Hemoglobin (Hb), Serum Ferritin (SF), Serum Transferrin Receptor (sTfR), and C - Reactive protein (CRP). Prevalence of iron deficiency anemia will be calculated based on the umber of subjects with Hb<115 g/l; SF<12 microgram/l.

SECONDARY OUTCOMES:
Serum Transferrin Receptor | 6 months, measurements will be done at start and at the end of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Abdul R Abizari, Msc, Principal Investigator — Division of Human Nutrition, Wageningen University
Locations (1):
- Department of Community Nutrition, University for Development Studies, Tamale, Ghana

REFERENCES:
- [Derived] Abizari AR, Moretti D, Zimmermann MB, Armar-Klemesu M, Brouwer ID. Whole cowpea meal fortified with NaFeEDTA reduces iron deficiency among Ghanaian school children in a malaria endemic area. J Nutr. 2012 Oct;142(10):1836-42. doi: 10.3945/jn.112.165753. Epub 2012 Aug 22. PMID 22915294